CLINICAL TRIAL: NCT07072572
Title: Lung Point Of Care Ultrasond (L-Pocus)-Guided Administration Of Intravenous Albumin In Decompensated Cirrhosis: A Pilot, Open Label, Randomized Controlled Trial
Brief Title: Lung Point of Care Ultrasound to Guide Albumin Administration in Cirrhosis
Acronym: POCUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centro Medico Issemym (Other)
Responsible Party: Principal Investigator, Luis Alejandro Rosales Renteria, Principal investigator, Centro Medico Issemym
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMedicoIssemym
Record Dates: First submitted 2025-04-20; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cirrhosis; Cirrhosis Advanced; Acute Kidney Injury; Ascites
Keywords: Albumin; Lung ultrasound
MeSH Terms: conditions — Fibrosis; Acute Kidney Injury; Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional albumin group (No Intervention): Conventional albumin group
- Lung ultrasound guided albumin administration group (Experimental): Lung ultrasound guided albumin administration group
  Interventions: Drug: Lower albumin dosage

INTERVENTIONS:
Drug: Lower albumin dosage — A fixed dose of 35 grams of albumin on they one and day two.
  Other Names: Lung ultrasound guided administration of albumin
  Arms: Lung ultrasound guided albumin administration group

SUMMARY:
To guide the administration of intravenous albumin by lung ultrasound in decompensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years.
* Decompensated cirrhosis
* Indication for intravenous albumin use

Exclusion Criteria:

* Development of variceal hemorrage before the administration of albumin, respiratory failure previous to albumin use, or the presence of hepatocellular carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Overall mortality at 30 days | 30 days
  Overall mortality at 30 days

SECONDARY OUTCOMES:
Respiratory failure | Every 24 hours, during hospitalization, (assesed up to 28 days)
  Number of Participants with respiratory failure, as defined as a requirement of greater than 10/L min og supplemental oxygen, a SpO2 lower than 92% on room temperature or an arterial blood oxyen concentration (pO2) lower than 60 mmHg.
Acute kidney injury | Every 24 hours, during hospitalization, (assesed up to 28 days)
  Number of Participants with acute kidney injury, as defined by the KDIGO criteria, being KDIGO 1 an increment in serum creatinine over baseline values of 0.3 mg/dL, KDIGO 2-2.9 times over baseline, KDIGO 3, 3 times over baseline.
Resolution of SBP | Day three of antibiotic treatment initiated for spontaneous bacterial peritonitis.
  Number of Participants with resolution of SBP: Defined as a reduction of 25% of WBC in ascites performed through check up paracentesis at day three.
Development of variceal hemorrhage | During hospitailization, (assesed up to 28 days)
  Number of Participants with development of variceal hemorrhage: Defined as upper GI bleeding due to gastroesophageal varices confirmed by endoscopy
acute-on-chronic liver failure | During hospitailization, (assesed up to 28 days)
  Number of Participants with development of acute on chronic liver failure, as defined by ther Ec-CLF criteria, which asses biochemical function of six organ systems: liver, kidney, brain, coagulation, circulation, and lungs. Each organ system is graded on a scale of 1 to 3, with higher scores indicating more severe organ dysfunction.
Total hospitalization time | 30 days
  Total hospitalization time

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Médico ISSEMyM, Metepec, State of Mexico, Mexico